CLINICAL TRIAL: NCT06642324
Title: Exploration of Human Papillomavirus Association and Genomic Characteristics in Head and Neck Squamous Cell Carcinomas in Bangladesh
Brief Title: Human Papillomavirus Association and Genomic Exploration in Head-Neck Squamous Cell Carcinomas
Acronym: HPV & HNSCC
Status: Recruiting | Type: Observational
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, S M Rashed Ul Islam, Associate Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Other Study IDs: BSMMU HNSCC Study-1
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Head Neck Cancer; Oropharyngeal Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms | interventions — Immunohistochemistry; Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biopsy sample, Mouth wash, whole blood, serum, paraffin embedded tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- HPV Positive HNSCC Population: Tissues from Head Neck Squamous Cell Carcinoma and HPV DNA-positive
  Interventions: Diagnostic Test: Histopathology, Immunohistochemistry, Real-Time PCR, Sequencing
- HPV Negative HNSCC Population: Tissues from Head Neck Squamous Cell Carcinoma and HPV DNA-negative
  Interventions: Diagnostic Test: Histopathology, Immunohistochemistry, Real-Time PCR, Sequencing
- Healthy Population: Healthy Population who does not have any carcinoma, chronic diseases, Genetic diseases, acute/chronic infectious diseases, etc.
  Interventions: Diagnostic Test: Histopathology, Immunohistochemistry, Real-Time PCR, Sequencing

INTERVENTIONS:
Diagnostic Test: Histopathology, Immunohistochemistry, Real-Time PCR, Sequencing — Histopathology for carcinoma detection, Immunohistochemistry for carcinoma-related protein expression, Real-Time PCR for HPV association and HPV typing, Sequencing for genetic study or mutation analysis.

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) represents a significant public health burden in Bangladesh with a high incidence and mortality rate. While traditional risk factors like tobacco and betel nut chewing contribute to HNSCC incidence, the emergence of HPV-associated HNSCC presents a unique challenge. The main goal of this observational study is to explore the prevalence, risk factors, and biological mechanisms underlying food habits and HPV-driven HNSCC in the population and identify the genomic changes and characteristics related to this malignancy. This study will provide the prevalence of HPV-associated HNSCC and screening the HPV typing in the Bangladeshi population, identify risk factors, and any biologically driven mechanisms causing HNSCC.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) represents Bangladesh's significant public health challenge. According to GLOBACAN data, these cancers are among the most prevalent malignancies in the country, with a considerable impact on morbidity and mortality rates. Several factors contribute to the high incidence of HNSCC in Bangladesh, including prevalent tobacco and betel nut chewing habits, poor oral hygiene practices, oncogenic viruses such as human papillomavirus (HPV), and limited access to healthcare facilities for early detection and treatment. In recent years, the incidence of HPV-associated HNSCC has been on the rise, posing a significant health concern globally. HPV16 and HPV18 have been strongly linked to the development of HNSCC. The global surge of HPV-associated HNSCC necessitates further investigation, particularly in regions like Bangladesh. By addressing these critical areas, this research has the potential to improve public health outcomes in Bangladesh significantly.

The main goal of this observational study is to explore the prevalence, risk factors, and biological mechanisms underlying food habits and HPV-driven HNSCC in the Bangladeshi population. Additionally, the study aims to identify the gene expression changes related to these factors.

At first, the HNSCC samples will be detected through histopathology analysis, followed by nucleic acid extraction from the carcinoma-positive samples. Subsequently, molecular screening will be conducted alongside an assessment of patient histories. Based on the results from the molecular screening, immunohistochemistry will be performed on both HPV-positive and HPV-negative HNSCC samples to assess carcinoma-related protein expression. Finally, a comprehensive cancer omics analysis will be conducted after obtaining the sequencing data. Understanding these aspects is crucial for developing targeted prevention strategies, including HPV vaccination campaigns and public health education initiatives on high-risk sexual behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Patient Age: adult (> 18 years)
2. Head and neck squamous cell carcinoma diagnosed by biopsy (Histopathology confirmed HNSCC).
3. Diagnosed cases specific Head-Neck sub-sites: (oral cavity, oropharynx, hypopharynx, larynx, tongue)
4. Patient's Consent

Exclusion Criteria:

1. Patient Age: children (< 18 years)
2. Cancers of any part of the body other than the head-neck region.
3. People without HNSCC
4. Any chronic diseases, genetic diseases, acute/chronic infectious diseases, etc. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A descriptive study will be conducted among head-neck squamous cell carcinoma people, who will be recruited after receiving informed written consent to participate. The study population will be recruited from the Department of Otolaryngology-Head & Neck Surgery, histopathology of the BSMMU, and laboratory work will be done at the Department of Virology, BSMMU. During the specimen collection, brief demographic and clinical data will be collected through a pre-designed written questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
HPV positivity in histopathological positive HNSCC detected tissue samples | 2 years
  To detect and type the HPV DNA in HNSCC tissue samples utilizing Real-Time PCR and Histopathology.

SECONDARY OUTCOMES:
Genetic predisposition to HNSCC due to virus, Food habit or Tobacco | 2 years
  To explore any influence of HPV positivity and food habits, like betel nut, betel leaf, tobacco, alcohol, etc, through genetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: S M Rashed Ul Islam, M. Phil, MPH, Principal Investigator — Bangabandhu Sheikh Mujib Medical University (BSMMU)
Locations (1):
- Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akhter M, Ali L, Hassan Z, Khan I. Association of human papilloma virus infection and oral squamous cell carcinoma in Bangladesh. J Health Popul Nutr. 2013 Mar;31(1):65-9. doi: 10.3329/jhpn.v31i1.14750. PMID 23617206
- [Background] Gao G, Wang J, Kasperbauer JL, Tombers NM, Teng F, Gou H, Zhao Y, Bao Z, Smith DI. Whole genome sequencing reveals complexity in both HPV sequences present and HPV integrations in HPV-positive oropharyngeal squamous cell carcinomas. BMC Cancer. 2019 Apr 11;19(1):352. doi: 10.1186/s12885-019-5536-1. PMID 30975103
- [Background] Lechner M, Frampton GM, Fenton T, Feber A, Palmer G, Jay A, Pillay N, Forster M, Cronin MT, Lipson D, Miller VA, Brennan TA, Henderson S, Vaz F, O'Flynn P, Kalavrezos N, Yelensky R, Beck S, Stephens PJ, Boshoff C. Targeted next-generation sequencing of head and neck squamous cell carcinoma identifies novel genetic alterations in HPV+ and HPV- tumors. Genome Med. 2013 May 29;5(5):49. doi: 10.1186/gm453. eCollection 2013. PMID 23718828
- [Background] Shaikh MH, Khan AI, Sadat A, Chowdhury AH, Jinnah SA, Gopalan V, Lam AK, Clarke DTW, McMillan NAJ, Johnson NW. Prevalence and types of high-risk human papillomaviruses in head and neck cancers from Bangladesh. BMC Cancer. 2017 Nov 25;17(1):792. doi: 10.1186/s12885-017-3789-0. PMID 29178862